CLINICAL TRIAL: NCT02823028
Title: Social Media Technology for Treating Tobacco Addiction
Brief Title: Twitter-enabled Mobile Messaging for Smoking Relapse Prevention (Tweet2Quit)
Acronym: Tweet2Quit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Stanford University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Cornelia Pechmann, Principle Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20141303; R01CA204356 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-07-06 (Estimated); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Smoking Cessation
Keywords: Smoking; Social Media; Twitter; Behavior Change; Social Support
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NRT + Web Guide (Active Comparator): NCI Smokefree.gov plus 8 weeks of combination NRT (nicotine patch plus gum/lozenges)
  Interventions: Drug: NRT; Behavioral: Web Guide
- NRT + Web Guide + Tweet2Quit-Coed (Experimental): NCI Smokefree.gov plus 8 weeks of combination NRT (nicotine patch plus gum/lozenges) plus assignment to a coed Tweet2Quit group
  Interventions: Drug: NRT; Behavioral: Web Guide; Behavioral: Tweet2Quit
- NRT + Web Guide + Tweet2Quit-Women (Experimental): Experimental: NRT + Web Guide + Tweet2Quit-Women NCI Smokefree.gov plus 8 weeks of combination NRT (nicotine patch plus gum/lozenges) plus assignment to a women-only Tweet2Quit group
  Interventions: Drug: NRT; Behavioral: Web Guide; Behavioral: Tweet2Quit
- Initial Pilot Group (NRT + Web Guide + Tweet2Quit-Coed) (Other): The initial pilot group was run to check technology functionality and user acceptance; it was not included in outcome assessments. These participants received NCI Smokefree.gov plus 8 weeks of combination NRT (nicotine patch plus gum/lozenges) plus assignment to a coed Tweet2Quit group.
  Interventions: Drug: NRT; Behavioral: Web Guide; Behavioral: Tweet2Quit

INTERVENTIONS:
Drug: NRT — 8-weeks of study provided NRT patch, and 8-weeks of study provided NRT gum of varying strengths or 8-weeks of study provided NRT lozenges, depending on patient level of nicotine dependence.
  Other Names: Nicotine Replacement Therapy
Behavioral: Web Guide — A website that will provide participants with access to an evidence-based set of "base" treatment materials in one central location. The site will include information on the proper use of nicotine patches, gum, lozenges, and it will have a direct link for participants to access the NCI's Smokefree.gov Quit Guide. The website will remind participants about quit dates and send alerts via email to participants to complete the appropriate NCI Quit Guide modules.
Behavioral: Tweet2Quit — A fully automated, 90-day quit smoking intervention that provides an online, peer-to-peer support group for quitting and uses twice-daily automessages to encourage and direct the peer-to-peer exchanges. Each group will consist of 12 buddy pairs (matched on key demographics) that will be introduced via automated texts. The program will generate twice-daily programmed contacts (e.g., "what benefits do you hope to get from quitting smoking?"). Automated pattern detection software will identify and address any problematic low tweeting within a group.
  Arms: Initial Pilot Group (NRT + Web Guide + Tweet2Quit-Coed); NRT + Web Guide + Tweet2Quit-Coed; NRT + Web Guide + Tweet2Quit-Women

SUMMARY:
Tweet2Quit is an innovative smoking cessation intervention that combines real-time online peer-to-peer support with auto messaging. In a three-group randomized controlled trial, the investigators will compare: 1) usual care, 2) Tweet2Quit-coed, and 3) Tweet2Quit-Women only.

DETAILED DESCRIPTION:
The proposed randomized controlled evaluation of the Tweet2Quit intervention will biochemically verify abstinence out to 6-months follow-up and will test the personalized benefit for women of a women-only versus co-ed Tweet2Quit group. In a 3-arm design, the investigators will compare: 1) usual care, 2) Tweet2Quit-coed, and 3) Tweet2Quit-Women only.

Each Tweet2Quit group will include buddy pairs based on similarity in demographics. Also automated pattern detection will identify dips in tweeting and trigger automated alerts and engagement strategies.

The sample consists of 960 adult smokers plus 20 in an initial pilot group to check technology functionality (not included in outcome assessment).

The primary aims test Hypothesis 1: Relative to usual care (n=240), Tweet2Quit-coed groups (n=480) will achieve significantly greater bioconfirmed sustained abstinence out to 6-months follow-up for each gender, and Hypothesis 2: Women in Tweet2Quit will achieve significantly greater bioconfirmed 6-months abstinence in woman-only groups (n=240) vs. coed groups (n=240 women).

Our secondary aims are to test the same hypotheses based on 3-month (end of treatment) sustained abstinence and 7-day point prevalence at 1, 3, and 6 months with biochemical verification at 3 and 6 months. Exploratory aims will study the Tweet2Quit groups' social network structures with a focus on the identification of buddy pairs and social brokers and test if these relationships are stronger for women in women-only groups versus women in coed groups of Tweet2Quit.

*Prior to the start of the RCT, the investigators will run one coed pilot group (N=20). Total size of the study (including the pilot group) will be N=980.

ELIGIBILITY:
Inclusion Criteria:

* Are 21-59 years of age
* Are smoking 5+ cigarettes/day and 100+ cigarettes in one's lifetime
* In the preparation stage of quitting smoking
* Are English speaking
* Have a mobile phone with an unlimited texting plan and internet access (via mobile phone)
* Text at least once a week
* Are a social media user
* Have an active email account
* Lives in the continental USA

Exclusion Criteria:

* Have certain medical conditions that are contraindicated for nicotine replacement therapy: pregnant, breast feeding, a recent heart attack, an irregular heartbeat, high blood pressure not controlled with medication, skin allergies to adhesive tape or serious skin problems, taking a prescription medicine for depression, and/or any other medical conditions that would prevent you from completing this study.
* Are an illicit hard drug user or regular marijuana user
* Share a household with someone else or has an immediate family member who has already enrolled in the study currently or in the past or if the participant has already been enrolled or failed to pass the screening once already since October 2016
* Participated in Tweet2Quit between 2012-2013 in a Twitter group and was not an active tweeter (<1 week)
* Fails to provide valid forms of all the required personal contact information

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 980 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie (Cornelia) Pechmann, PhD, MBA, MS, Principal Investigator — University of California, Irvine; Judith J Prochaska, PhD, MPH, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California, Irvine - Paul Merage School of Business, Irvine, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pechmann C, Phillips C, Calder D, Prochaska JJ. Facebook Recruitment Using Zip Codes to Improve Diversity in Health Research: Longitudinal Observational Study. J Med Internet Res. 2020 Jun 5;22(6):e17554. doi: 10.2196/17554. PMID 32501274
- [Derived] Pechmann CA, Calder D, Phillips C, Delucchi K, Prochaska JJ. The Use of Web-Based Support Groups Versus Usual Quit-Smoking Care for Men and Women Aged 21-59 Years: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jan 14;9(1):e16417. doi: 10.2196/16417. PMID 31934869
- See also: Please visit the Tweet2Quit Website to apply! — http://tweet2quit.merage.uci.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled in the coed pilot group arm (N=20), as preplanned, were not contacted for follow-up assessments. The pilot group arm was included solely to test the technical setup of the online support groups, e.g., to make sure the automated messaging and automated buddy pairing were working properly. The pilot group arm was never intended to be included in the outcome assessments.
Groups:
- Coed Pilot Group Arm: Technical setup of online support groups only.
Period: Overall Study
Arm/Group | NRT + Web Guide | NRT + Web Guide + Tweet2Quit-Coed | NRT + Web Guide + Tweet2Quit-Women | Coed Pilot Group Arm
Started | 240 | 480 | 240 | 20
Completed | 235 | 457 | 230 | 20
Not Completed | 5 | 23 | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot: A coed pilot group was run to test the support groups functionality only. Outcome measures were not obtained on the coed pilot group; only baseline measures were obtained.
- Total: Total of all reporting groups
Arm/Group | NRT + Web Guide | NRT + Web Guide + Tweet2Quit-Coed | NRT + Web Guide + Tweet2Quit-Women | Pilot | Total
Number analyzed (Participants) | 240 | 480 | 240 | 20 | 980
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 240 | 480 | 240 | 20 | 980
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.37 (9.685) | 39.04 (9.524) | 39.75 (9.450) | 39 (9) | 39.55 (9.552)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 338 | 240 | 14 | 759
  Male | 73 | 142 | 0 | 6 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 21 | 6 | 2 | 39
  Not Hispanic or Latino | 228 | 454 | 232 | 18 | 932
  Unknown or Not Reported | 2 | 5 | 2 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 1 | 0 | 10
  Asian | 3 | 5 | 2 | 0 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 21 | 55 | 22 | 2 | 100
  White | 207 | 397 | 210 | 18 | 832
  More than one race | 2 | 13 | 2 | 0 | 17
  Unknown or Not Reported | 2 | 5 | 3 | 0 | 10
Region of Enrollment [Number; unit: participants]
  United States | 240 | 480 | 240 | 20 | 980
Cigarettes/Day [Mean (Standard Deviation); unit: cigarettes/day] | 17.8 (8.4) | 17.3 (7.7) | 17.8 (7.2) | 17 (8) | 17.6 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 6-month Sustained Abstinence
Description: Percentage of participants who reported no use of tobacco products by answering the questions: 'How many cigarettes have you smoked', 'How many other tobacco products have you used', and 'How many times have you used e-cigs' since the quit date (assessed at 1, 3 and 6 months post quit date) confirmed by salivary cotinine measurement (assessed at 3 and 6 months post quit date). Note: We will apply the Russell Standard for abstinence, allowing 5 or fewer instances of tobacco use over 6 months.
  In our primary (most rigorous) analysis, we will consider a cotinine-positive test, regardless of source, to be non-abstinent. In additional analyses, we will code as abstinent those who assert tobacco abstinence but continue use of FDA-approved nicotine replacement therapy. In other analyses we will report results with ENDS-only users coded first as non-abstinent and then for comparison as abstinent.
Time Frame: 6 Month
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Web Guide | NRT + Web Guide + Tweet2Quit-Coed | NRT + Web Guide + Tweet2Quit-Women
Number analyzed (Participants) | 235 | 457 | 230
Participants | 23 | 45 | 18
Statistical Analysis 1: Comparison: NRT + Web Guide vs NRT + Web Guide + Tweet2Quit-Women; Test type: Superiority; p = .779, Chi-squared; Odds Ratio (OR) = .931

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | NRT + Web Guide | NRT + Web Guide + Tweet2Quit-Coed | NRT + Web Guide + Tweet2Quit-Women | Pilot
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/480 | 0/240 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/480 | 0/240 | 0/20
Other Adverse Events (participants affected / at risk) | 0/240 | 0/480 | 0/240 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02823028/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02823028/SAP_001.pdf